CLINICAL TRIAL: NCT01490177
Title: Single Center, Phase I Food Allergy Oral Immunotherapy Study
Brief Title: Single Center Food Allergy Oral Immunotherapy Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kari Christine Nadeau, Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22871
Record Dates: First submitted 2011-11-29; First posted 2011-12-12 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Immune System Diseases
Keywords: Multiple food allergies
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- One (Experimental)
  Interventions: Drug: Food proteins

INTERVENTIONS:
Drug: Food proteins — Oral ingestion of Food proteins

SUMMARY:
The Primary Objective of the study is to develop a customized regimen for oral immunotherapy that reflects what the subject is allergic in a clinically significant way (i.e., the offending food allergen is defined as a food allergen with a positive skin test or positive specific IgE and a positive DBPCFC). Therefore, the investigators prefer that both single and multiple food allergy subjects are included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe peanut and/or egg and/or milk and/or tree nut and/or seed allergic subjects between the ages of 4 to 55 years old.
* Sensitivity to food allergen will be documented by a positive skin prick test result (see Appendix for details) or allergen specific ImmunoCAP IgE level with 7 kU/L as a lower limit of eligibility.

Exclusion Criteria:

* No absolute contraindications are known. However, the risk of serious systemic anaphylactic reactions to food allergens suggests a number of preexisting conditions that should be considered relative contraindications. Among those conditions are acute infections, autoimmune disease, severe cardiac disease, and treatment with beta-adrenergic antagonistic drugs (beta-blockers).
* Subjects having a history of severe anaphylaxis to food allergens that will be desensitized in this study requiring intubation or admission to an ICU, frequent allergic or non-allergic urticaria, or history consistent with poorly controlled persistent asthma.

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of adverse events in the treatment population | 2 years

SECONDARY OUTCOMES:
Number of subjects who reach 2g or more of food flour | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Begin P, Winterroth LC, Dominguez T, Wilson SP, Bacal L, Mehrotra A, Kausch B, Trela A, Hoyte E, O'Riordan G, Seki S, Blakemore A, Woch M, Hamilton RG, Nadeau KC. Safety and feasibility of oral immunotherapy to multiple allergens for food allergy. Allergy Asthma Clin Immunol. 2014 Jan 15;10(1):1. doi: 10.1186/1710-1492-10-1. PMID 24428859